CLINICAL TRIAL: NCT04203992
Title: TRUE CHAMPION: An Educational Videogame Intervention for the Prevention of Doping and Supplement Abuse in Teenage Athletes
Brief Title: Videogame for the Prevention of Doping and Supplement Abuse in Teenage Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University (Other)
Collaborators: International Olympic Committee (Unknown); World Anti-Doping Agency (Other); Phantom Compass (Unknown); Digitalmill, Inc. (Unknown)
Responsible Party: Principal Investigator, Lindsay Duncan, Associate Professor, William Dawson Scholar, McGill University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 476-0418
Record Dates: First submitted 2019-12-11; First posted 2019-12-18 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Doping in Sport; Performance Enhancing Product Use
Keywords: Student athletes; Supplements; Videogame

STUDY DESIGN:
Intervention Model Description: We aim to enroll 284 male and female student-athletes between the ages of 13 and 16. Participants will be assigned to either an intervention group (n = 142) or a comparison group (n = 142).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Videogame (Experimental): Educational videogame, five 60-minute sessions over one month
  Interventions: Behavioral: Videogame
- Booklet (Active Comparator): Educational booklet, one session
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Videogame — True Champion is an educational, values-based game that aims to empower young athletes to make informed decisions to avoid doping.
  Participants engaging in the videogame sessions will encounter a series of thought-provoking situations and knowledge tests. Players will help their assigned character navigate through these curriculum-rich scenarios in order to reach their performance goals in a healthy and ethical way.
  Arms: Videogame
Behavioral: Control — Participants will be given an anti-doping booklet prepared by UNESCO. This booklet is considered standard educational material, i.e. what might be presented to young athletes as part of their regular sports curriculum.
  Arms: Booklet

SUMMARY:
The purpose of this research is to test the effectiveness of an interactive doping education videogame among student athletes. Specifically, the game will teach athletes aged 13-16 years about the risks of doping and will foster the values, motivation, and behavioural skills needed to avoid temptation and pressure to dope. The investigators hypothesize that student athletes who play the intervention game will have lower use of banned substances and sport supplements, greater intentions to stay clean, and will also show improvements in the cognitive and motivational antecedents to doping when compared to a control condition.

DETAILED DESCRIPTION:
284 student athletes will be enrolled in this two-arm quasi-experimental study. The participants will be boys and girls, aged 13 to 16 years who compete in any sport. Participants will be recruited and enrolled through partnerships with their school physical education and/or sport programs. Participants will complete baseline questionnaires assessing demographics, history of sport participation, and psychological variables related to doping prevention including knowledge, doping self-regulatory efficacy, motivation, attitudes, intentions, perceived norms, doping refusal, substance use behaviours, and doping related protective behaviours (e.g., checking the list of ingredients on medications). Participants will then be assigned to either an intervention group (n = 142; the doping videogame the investigators are developing) or a comparison group (n = 142). The comparison group will be given printed educational materials about doping education, developed by an accredited source (e.g., UNESCO). Assignment to the intervention or comparison group will be conducted at the level of the school to reduce the potential for contamination that could occur if intervention and comparison students were interacting in their school environment and sharing information they learned from the game. Participants from the intervention group will play five, 60-minute sessions over the course of one month (5 hours of total gameplay). Before the gameplay sessions begin, the Project Director and research assistants will orient the intervention group participants to the use of the intervention videogame. Players will be given a tutorial on an iPad demonstrating the mechanics of the game and how to use the iPad. Each player will have their own dedicated iPad that they will use during each game play session (this will be provided by the research team). Shortly after the last gameplay session is completed, participants from both groups will be asked to complete a questionnaire assessing the same psychological variables assessed at baseline as well as their gameplay experience. The psychological variables will also be assessed at three, six, and 12 month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Subject competes in a competitive sport at the high school level or higher
* Able to read and understand English

Exclusion Criteria:

* None

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 284 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Use of banned substances | 12 months
  Self-reported use of banned substances for performance enhancement or recovery in sport.
  This outcome will be measured using a self-reported questionnaire.
  Scale: Performance-Enhancing Substances and Methods Use
  Minimum value: 1 - extremely unlikely (better outcome)
  Maximum value: 7 - extremely likely (worse outcome)
Use of sport supplements | 12 months
  Self-reported use of supplements for performance enhancement or recovery in sport.
  This outcome will be measured using a self-reported questionnaire.
  Scale: Performance-Enhancing Substances and Methods Use
  Minimum value: 1 - extremely unlikely (better outcome)
  Maximum value: 7 - extremely likely (worse outcome)
Intentions to use banned substances and sport supplements | 12 months
  Self-reported intentions of using banned substances or supplements for performance enhancement or recovery in sport.
  This outcome will be measured using a self-reported questionnaire.
  Scale: Performance-Enhancing Substances and Methods Use
  Minimum value: 1 - extremely unlikely (better outcome)
  Maximum value: 7 - extremely likely (worse outcome)

SECONDARY OUTCOMES:
Knowledge | 12 months
  Knowledge of anti-doping rules, definitions and consequences of doping.
  This outcome will be assessed using a True/False questionnaire.
Doping Self-Regulatory Efficacy | 12 months
  Self-efficacy for refusing doping under a variety of pressure situations.
  This outcome will be measured using a validated questionnaire.
  Scale: Doping Self-Regulatory Efficacy
  Minimum value: 1 - no confidence (better outcome)
  Maximum value: 5 - complete confidence (worse outcome)
Motivation | 12 months
  Motivations for abstaining from doping.
  This outcome will be measured using an adaptation of a validated questionnaire.
  Scale: Treatment Self-Regulation Questionnaire for the Avoidance of Doping in Sport
  Minimum value: 1 - not true at all (worse outcome)
  Maximum value: 7 - very true (better outcome)
Attitudes | 12 months
  Attitudes towards doping in sport.
  This outcome will be measured using a subscale from a validated questionnaire.
  Scale: The Adolescent Sport Doping Inventory
  Minimum value: 1 - strongly disagree (worse outcome)
  Maximum value: 7 - strongly agree (better outcome)
  Note: some items are reverse-scored
Anti-doping protective behaviours | 12 months
  Self-reported engagement in behaviours linked to doping abstinence.
  Scale: Microbehaviours
  Minimum value: 1 - never (worse outcome)
  Maximum value: 7 - always (better outcome)
Doping refusal | 12 months
  Self-report of having refused a supplement or performance-enhancing substance.
  This outcome will be assessed using a Yes (worse outcome) or No (better outcome) questionnaire.
Gameplay experience | 1 month
  Enjoyment and acceptability of the True Champion videogame among players assigned to the intervention condition.
  This outcome will be assessed using a questionnaire we have created. Answers will range from "strongly disagree" to "strongly agree".

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay R Duncan, PhD, Principal Investigator — McGill University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goulet C, Valois P, Buist A, Cote M. Predictors of the use of performance-enhancing substances by young athletes. Clin J Sport Med. 2010 Jul;20(4):243-8. doi: 10.1097/JSM.0b013e3181e0b935. PMID 20606508
- [Background] Boardley I, Smith AL, Mills JP, Grix J, Wynne C., & Wilkins L. Development of Moral Disengagement and Self-Regulatory Efficacy Assessments Relevant to Doping in Sport and Exercise. SportRxiv, 12 Oct. 2017. Web.
- [Background] Chan DK, Dimmock JA, Donovan RJ, Hardcastle S, Lentillon-Kaestner V, Hagger MS. Self-determined motivation in sport predicts anti-doping motivation and intention: a perspective from the trans-contextual model. J Sci Med Sport. 2015 May;18(3):315-22. doi: 10.1016/j.jsams.2014.04.001. Epub 2014 Apr 13. PMID 24793786
- [Background] Nicholls AR, Levy AR, Meir R, Sanctuary C, Jones L, Baghurst T, Thompson MA, Perry JL. The development and validation of the Adolescent Sport Drug Inventory (ASDI) among athletes from four continents. Psychol Assess. 2019 Nov;31(11):1279-1293. doi: 10.1037/pas0000750. Epub 2019 Jul 18. PMID 31318254